CLINICAL TRIAL: NCT06807619
Title: BrainMet ADePPT (Anticancer Drug Penetration Platform Trial)
Brief Title: A Study of Sotorasib in People With Brain Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-111
Record Dates: First submitted 2025-01-29; First posted 2025-02-04 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Brain Tumor
Keywords: SOTORASIB; KRAS G12C; CNS-BRAIN; Advanced; 24-111
MeSH Terms: conditions — Brain Neoplasms | interventions — sotorasib

STUDY DESIGN:
Intervention Model Description: Patients will be separated into cohorts based on wether they are drug/combination of interest (DCOInaïve) or have progressed on the DCOI.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- DCOI naïve (Experimental): Will receive the standard dose of sotorasib.
  Interventions: Drug: Sotorasib
- Progressed on the DCOI (Active Comparator): Will continue to receive the sotorasib dose they were previously receiving, according to their doctor's instruction.
  Interventions: Drug: Sotorasib

INTERVENTIONS:
Drug: Sotorasib — Enrolled patients will be administered DCOI at the FDA-recommended dose or continued on the DCOI at the discretion of the treating Oncologist per standard of care
  Other Names: AMG 510

SUMMARY:
The researchers are doing this study to find out how effective sotorasib is at getting into KRAS G12C+ brain tumors. The researchers will also find out whether sotorasib is a safe and effective treatment for people undergoing surgical resection of KRAS G12C+ metastatic brain tumors, and do tests that show how the body absorbs, distributes, and gets rid of sotorasib.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 18 years of age with one or more brain tumors planned for neurosurgical resection/biopsy
* Patients with concomitant leptomeningeal metastasis are eligible provided they have parenchymal brain neoplastic disease requiring resection/biopsy
* For all cohorts: no limit on prior CNS radiation or systemic therapyKPS ≥ 60
* Life expectancy >12 weeks
* Adequate treatment washout period from prior therapies to allow recovery from any prior treatment-related toxicities before enrollment in the judgment of the Investigator
* Adequate bone marrow, renal, hepatic, and coagulation parameters (obtained ≤7 days prior to the first day of study treatment):

  * Absolute neutrophil count (ANC) ≥1.0 × 10^3/μL (granulocyte-colony stimulating factor administration is not allowed within 1 week prior to C1D1)
  * Platelet count ≥10.0x10^4/μL. Note: Participants requiring ongoing transfusions or growth factor support to maintain platelet count ≥10.0x10^4/μL are not eligible. (Platelet transfusion is not allowed within 1 week prior to C1D1)
  * Hemoglobin ≥ 7.0 g/dL (≥ 8 g/dL in gastric cancer / gastroesophageal cancer indications). Note: Participants requiring ongoing transfusions or growth factor support to maintain hemoglobin ≥8.0 g/dL are not eligible (Red blood cell transfusion is not allowed within 1 week prior to C1D1)
  * Creatinine clearance ≥30 mL/min, as calculated using the Cockcroft-Gault equation
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤3 × upper limit of normal (ULN) (<5x ULN in participants with liver metastases)
  * Total bilirubin ≤1.5 × ULN) if no liver metastases or <3 × ULN in the presence of documented Gilbert's syndrome (unconjugated hyperbilirubinemia) or liver metastases at baseline

Exclusion Criteria:

* Known allergy or hypersensitivity to study treatment or any of the study drug excipients. For patients who are allergic to gadolinium-based agents may receive premedication as per institutional protocol or imaged without contrast at the discretion of the Principal Investigator; reactions will be managed per standard institutional protocol
* Multiple primary malignancies within 3 years, with the exception of:

  * adequately resected non-melanoma skin cancer
  * carcinoma in situ of the cervix
  * Smoldering pre-malignant or malignant conditions with minimal concern for CNS or extracranial progression during treatment such as CLL or MGUS based on the assessment of the treating provider
  * curatively treated in-situ disease
  * other solid tumors curatively treated
  * for patients with metastatic breast cancer: contralateral breast cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-01-29 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
ORR (overall response rate) | 1 year
  defined as the sum of CR (complete response) rate plus PR (partial response) rate, assessed by RECIST 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Nelson Moss, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering at Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Suffolk- Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering West Harrison (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm